CLINICAL TRIAL: NCT04447027
Title: A Phase 1 Study of Romidepsin, CC-486 (5-azacitidine), Dexamethasone, and Lenalidomide (RAdR) for Relapsed/Refractory T-cell Malignancies
Brief Title: Romidepsin, CC-486 (5-azacitidine), Dexamethasone, and Lenalidomide (RAdR) for Relapsed/Refractory T-cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Max Gordon, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200127; 20-C-0127
Record Dates: First submitted 2020-06-24; First posted 2020-06-25 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cutaneous T-Cell Lymphoma; Mature T-cell Malignancies; Peripheral T-Cell Lymphoma; Relapsed/ Refractory T-cell Malignancies
Keywords: Immunomodulatory Drugs (IMiDs); TCM; ALCL; Histone Deacetylase Inhibitors (HDACi)
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral | interventions — romidepsin; Lenalidomide; cc-486; Dexamethasone; Azacitidine; Electrocardiography; Biopsy; Magnetic Resonance Imaging; Spinal Puncture; Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1- Experimental Treatment: Dose Escalation (Experimental): Lenalidomide by oral intake at escalating doses of 5, 10, 15, or 20 mg/day on days -7 to 10 of each 21-day cycle (max 6 cycles) with CC-486 (5-azacitidine) at 300mg/day by oral intake on days 1-10, romidepsin at 12mg/m^2 by intravenous (IV) infusion on Day 1 and 10 and dexamethasone at 40mg by oral intake on days 1 and 10 of each cycle, to determine maximum tolerated dose (MTD).
  Interventions: Drug: Romidepsin; Drug: Lenalidomide; Drug: CC-486 (5-azacitidine); Drug: Dexamethasone; Diagnostic Test: EKG; Procedure: Bone Marrow Aspiration/Biopsy; Diagnostic Test: MRI; Procedure: Lumbar Puncture; Diagnostic Test: TTE
- 2 - Experimental Treatment: Dose Expansion (Experimental): Lenalidomide by oral intake at maximum tolerated dose (MTD) on days -7 to 10 of each 21-day cycle (max 6 cycles) with CC-486 (5-azacitidine) at 300mg/day by oral intake on days 1-10, romidepsin at 12mg/m^2 by intravenous (IV) infusion on Day 1 and 10 and dexamethasone at 40mg by oral intake on days 1 and 10 of each cycle
  Interventions: Drug: Romidepsin; Drug: Lenalidomide; Drug: CC-486 (5-azacitidine); Drug: Dexamethasone; Diagnostic Test: EKG; Procedure: Bone Marrow Aspiration/Biopsy; Diagnostic Test: MRI; Procedure: Lumbar Puncture; Diagnostic Test: TTE

INTERVENTIONS:
Drug: Romidepsin — Romidepsin (12mg/ m^2) will be administered on days 1 and 10 of each cycle through a peripheral or central intravenous catheter for 6 cycles.
  Other Names: Istodax
Drug: Lenalidomide — Lenalidomide will be administered by oral intake in a dose-escalation with a starting dose of 5mg daily, a second dose level of 10mg daily, a third dose level at 15mg daily, and a fourth dose level at 20mg daily on days -7 to day 10 of first cycle. After the second cycle, lenalidomide will be given from day 1 to day 10 in each cycle for up to 6 cycles.
  Other Names: REVLIMID
Drug: CC-486 (5-azacitidine) — CC-486 (5-azacitidine) with a dose of 300mg oral intake daily will be given on day 1 to day 10 for 6 cycles.
  Other Names: ONUREG
Drug: Dexamethasone — Dexamethasone, 40mg, by mouth (PO), will be given on days 1 and 10 of each cycle.
  Other Names: azacitidine tablets
Diagnostic Test: EKG — Screening
  Other Names: Electrocardiogram
Procedure: Bone Marrow Aspiration/Biopsy — Baseline, end of treatment and disease progression, and Day 30 (+7).
  Other Names: BM Aspiration/Bx
Diagnostic Test: MRI — Baseline, every 2 cycles, end of treatment and disease progression, and follow-up.
  Other Names: Magnetic resonance imaging
Procedure: Lumbar Puncture — Baseline, every 2 cycles, end of treatment and disease progression, and follow-up.
  Other Names: LP
Diagnostic Test: TTE — Screening
  Other Names: Transthoracic echocardiogram

SUMMARY:
Background:

Mature T-cell malignancies (TCMs) are a rare group of cancers that usually do not have effective treatments or cures. Because of this, participants with TCMs often relapse and have a poor overall prognosis. This trial is testing if combining several drugs against TCMs can be a more effective.

Primary Objective:

To test if the combination of romidepsin, CC-486 (5-azacitidine), dexamethasone, and lenalidomide (RAdR) can be given safely to participants with relapsed or treatment refractory TCM.

Other (Secondary) Objective:

Measure the activity of this combination treatment.

Eligibility:

People age 18 and older who have a failed or relapsed after standard treatments for mature TCMs.

Design:

Participants will be screened for eligibility by performing the following tests or procedures:

Physical exam

Medical history

Medicine review

Blood and urine tests

Symptom review

Bone marrow examination

Total Body imaging scans or x-rays

Tumor biopsy

Participants will have blood tests during treatment to make sure their blood cell counts are okay.

Romidepsin is infused through an intravenous (IV) placed in one of the veins usually in the arm. Lenalidomide, dexamethasone, and CC-486 (5-azacitidine) are pills or capsules taken by mouth.

Participants are asked to keep a diary of when they take their pills to make sure they are taking these medicines properly.

Participants will have tumor imaging scans after every 2nd cycle (or 6 weeks) to check if the treatment is working. If the doctors are concerned the cancer has spread to the brain and/or spine, they will have scans of the area(s) and a sampling of the fluid around the brain/spine which is obtained through a small needle inserted into the lower part of the back for a short time to collect the fluid. This procedure is called a spinal tap or lumbar puncture.

Participants who have tumor in their skin will have repeat exams of their skin and sometimes photographs taken of these areas to see if the treatment is working.

Participants will also be asked to give blood, saliva, and sometimes have optional biopsies of their tumor where these tests are done for research purposes.

After they have completed the protocol treatment (6 cycles), they will be asked to return to clinic 30 days after treatment has ended, then every other month (or 60 days) for the first 6 months, then every 3 months (90 days) for 2 years, and then every 6 months for years 2 to 4 after completing treatment. After 4.5 years, they will be seen once a year.

DETAILED DESCRIPTION:
Background:

* Mature T-cell malignancies (TCM) are rare and heterogeneous group of leukemias and lymphomas accounting for 5 to 10% of all lymphomas in the US
* Patients with systemic TCM are most commonly treated with a CHOP (cyclophosphamide, doxorubicin, vincristine and prednisone)-like regimens, that produce long-term progression-free survival in about 30% of these cases
* Patients with relapsed/refractory (R/R) TCM have very poor prognosis with median overall survival of less than 1 year. Treatment options for R/R TCM are very few and of limited efficacy, thus novel treatment strategies are urgently needed.
* Mutations in epigenetic regulators are common in aggressive TCMs and standard treatment with histone deacetylase inhibitors (HDACi) such as romidepsin show modest clinical activity with single agent the overall response (ORR) around 25%
* Combination of romidepsin and 5-azacitidine (hypomethylating agents) was synergistic in preclinical models, and has demonstrated high clinical activity with an ORR of 79%
* Many TCMs rely on The Ikaros-dependent nuclear factor κB (NF-κB)/interferon regulatory factor 4 (IRF4) signaling pathway to maintain proliferation, which is why lenalidomide, which induces degradation of Ikaros and downregulates IRF4, has single agent activity in R/R TCM with overall response rate (ORR) of 26% to 42%, depending on the subtype.
* Lenalidomide synergizes with romidepsin and enhances tumor cell death in TCM cell lines, predicting that the addition of lenalidomide to the established romidepsin/ CC-486 (5-azacitidine) combination will further improve efficacy.

Objectives:

-To determine the safety and toxicity profile and the maximum tolerated dose (MTD) of the four-drug combination of CC-486 (5-azacitidine), romidepsin, lenalidomide and dexamethasone in patients with TCM

Eligibility:

* Refractory/relapsed TCM (excluding in Cutaneous T-Cell Lymphoma) defined as follows:

  * Patients with systemic disease
  * Have received at least one line of prior therapy
  * Must have received brentuximab vedotin if the disease is anaplastic large cell lymphoma or cluster of differentiation 30 (CD30)-positive cutaneous T-cell lymphoma
* Age >= 18 years of age
* Eastern Cooperative Oncology Group performance status of <= 2 (or <= 3 if decrease is due to the disease)
* Histologically or cytologically confirmed relapsed and/or refractory mature TCM
* Adequate organ and marrow function

Design:

* Open-label, single-center, uncontrolled Phase 1 study
* 3 + 3 design will be used to determine the maximum tolerated dose (MTD) of dose-escalated lenalidomide with fixed dose of romidepsin and CC-486 (5-azacitidine)
* An expansion cohort of 9 patients will be evaluated at the MTD
* Maximum 6 cycles (28-day cycle) of combination therapy
* To explore all dose levels, including further evaluation in a dose expansion cohort, the accrual ceiling will be set at 30 patients

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have relapsed after or progressed during at least one line of prior systemic therapy (which may include allogeneic stem cell transplantation) for mature T or NK/T neoplasm, i.e. have relapsed and/or refractory mature T and natural killer (NK) neoplasm per 2016 World Health Organization (WHO) classification excluding chronic lymphoproliferative disorder of NK cells, aggressive NK-cell leukemia, and Cutaneous T-Cell Lymphoma.
* T or NK/T neoplasm from initial diagnosis or recurrence must be histologically or cytologically proven and diagnosis be confirmed by the Laboratory of Pathology, National Cancer Institute (NCI),
* Patients with anaplastic large cell lymphoma (ALCL) or cluster of differentiation (CD30) positive mycosis fungoides (MF) or Sézary syndrome (SS) must have relapsed after or become intolerant to prior anti-CD30 targeting therapy treatment with brentuximab vedotin
* For patients without circulating leukemia/lymphoma cells detectable by flow cytometry, a formalin fixed tissue block or 15 slides of tumor sample (archival or fresh) must be available at enrollment for performance of correlative studies. NOTE: Patients without circulating malignant cells must be willing to have a tumor biopsy if prior tissue or adequate archival tissue is not available (i.e., post-enrollment and prior to treatment).
* Disease must be measurable with at least one measurable lesion by response evaluation criteria in lymphoma (RECIL) 2017 or Modified Severity-Weighted Assessment Tool (mSWAT) criteria, or have an abnormal clonal T-cell population detectable by peripheral blood flow cytometry
* Age >18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <=2, or <= 3 if the decreased performance status is deemed to be due to disease and not residual toxicity from prior therapy or other causes.
* Adequate organ and marrow function as defined below:

  * Absolute neutrophil count >= 1,000/mcL
  * Platelets >= 75,000/mcL
  * Total bilirubin <= 1.5 X institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) <= 2.5 X institutional upper limit of normal (ULN)
  * Serum Creatinine <= 1.5 mg/dL OR
  * Creatinine Clearance >= 60 mL/min/1.73 m^2 as calculated by direct measurement of 24-hour urine for creatinine clearance
* Negative serum or urine pregnancy test at screening for women of childbearing potential (WOCBP) NOTE: WOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal. WOCBP must have a negative pregnancy test (hemoglobin (HCG) blood or urine) during screening.
* All study participants must be registered into the mandatory Revlimid REMS(R) program and be willing and able to comply with the requirements of the Risk Evaluation and Mitigation Strategy (REMS(R) program.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 6 months after completion of treatment for women, and for at least 3 months after completion of treatment for men. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS(R) program.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Anti-cancer treatment within 2 weeks prior to enrollment. (4 weeks for monoclonal antibodies and 6 weeks for nitrosoureas or mitomycin C).
* Patients who have received two of the following drugs at any point: lenalidomide, romidepsin, and 5-azacitidine. Patients who have received only one of the three drugs remain eligible.
* Patients with a diagnosis of cutaneous T-cell lymphoma (CTCL) are excluded from participation in the expansion cohort.
* Other malignancy that requires ongoing systemic hormonal therapy, chemotherapy, or immunotherapy.
* History of allergic reactions or known or suspected hypersensitivity attributed to compounds of similar chemical or biologic composition to lenalidomide, romidepsin and 5-azacitidine
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring systemic therapy, or psychiatric illness/social situations that would limit compliance with study requirements.
* Human immunodeficiency virus (HIV)-infected patients on effective antiretroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* History of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), celiac disease (i.e., sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the study drug and/or predispose the subject to an increased risk of gastrointestinal toxicity.
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (>= New York Heart Association Classification Class II), congenital long QT syndrome, or other serious cardiac arrhythmia including 2nd degree atrio ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min).
* Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes.
* Uncontrolled hypertension, i.e., blood pressure (BP) of >=160/95; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria.
* Triplicate average baseline QT corrected for heart rate by Fridericia's (QTcF) interval >= 480 ms
* Patients taking drugs leading to significant QT prolongation Note: A 5 half-life washout period must have elapsed following the use of these drugs prior to administration of romidepsin.
* Concomitant use of rifampin and other strong cytochrome P450 3A4 (CYP3A4) inhibitors and inducers within 2 weeks prior to starting protocol therapy.
* Other severe acute or chronic medical conditions including psychiatric conditions such as recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Pregnant or lactating women. Pregnant women are excluded from this study because lenalidomide is a Class X agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lenalidomide, breastfeeding should be discontinued if the mother is treated with lenalidomide. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Max Gordon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely. Genomic data will be available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data will be made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0127.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide: T-cell Malignancies, Dose Escalation, Arm 1, Dose Level -1
  Arm 1, Dose Level -1: Lenalidomide 2.5 mg Day 1-10 (7 days lead in for first cycle); CC-486 (5azacitidine) 200 mg by mouth (PO Day) 1 to 10; Romidepsin 12 mg/m^2 intravenous (IV) Day 1 and day 10; Dexamethasone 40 mg PO Day 1 and day 10. Relapsed/refractory mature T cell malignancies for determination of maximum tolerated dose (MTD).
- Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide: T-cell Malignancies, Dose Escalation, Arm 1, Dose Level 1
  Arm 1, Dose Level 1: Lenalidomide 5 mg Day 1-10 (7 days lead in for first cycle); CC-486 (5azacitidine) 300 mg by mouth (PO Day) 1 to 10; Romidepsin 12 mg/m^2 intravenous (IV) Day 1 and day 10; Dexamethasone 40 mg PO Day 1 and day 10. Relapsed/refractory mature T cell malignancies for determination of maximum tolerated dose (MTD).
- Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide: T-cell Malignancies, Dose Escalation, Arm 1, Dose Level 2
  Arm 1, Dose Level 2: Lenalidomide 10 mg Day 1-10 (7 days lead in for first cycle); CC-486 (5azacitidine) 300 mg by mouth (PO Day) 1 to 10; Romidepsin 12 mg/m^2 intravenous (IV) Day 1 and day 10; Dexamethasone 40 mg PO Day 1 and day 10. Relapsed/refractory mature T cell malignancies for determination of maximum tolerated dose (MTD).
- Arm 1, Cohort 1, Dose Level 3 Dose Escalation: T-cell Malignancies, Dose Escalation, Arm 1, Dose Level 3
  Arm 1, Dose Level 3: Lenalidomide 15 mg Day 1-10 (7 days lead in for first cycle); CC-486 (5azacitidine) 300 mg by mouth (PO Day) 1 to 10; Romidepsin 12 mg/m^2 intravenous (IV) Day 1 and day 10; Dexamethasone 40 mg PO Day 1 and day 10. Relapsed/refractory mature T cell malignancies for determination of maximum tolerated dose (MTD).
- Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide: T-cell Malignancies, Dose Escalation, Arm 1, Dose Level 4
  Arm 1, Dose Level 4: Lenalidomide 20 mg Day 1-10 (7 days lead in for first cycle); CC-486 (5azacitidine) 300 mg by mouth (PO Day) 1 to 10; Romidepsin 12 mg/m^2 intravenous (IV) Day 1 and day 10; Dexamethasone 40 mg PO Day 1 and day 10. Relapsed/refractory mature T cell malignancies for determination of maximum tolerated dose (MTD).
- Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide: T-cell Malignancies, Dose Expansion, Arm 2, Dose Level 2
  Arm 2, Dose Level 2: Lenalidomide by oral intake at maximum tolerated dose (MTD) on days -7 to 10 of each 21-day cycle (max 6 cycles) with CC-486 (5-azacitidine) at 300mg/day by oral intake on days 1-10, Romidepsin at 12 mg/m^2 by intravenous (IV) infusion on Day 1 and day 10; and Dexamethasone at 40 mg by oral intake on days 1 and 10 of each cycle. Relapsed/refractory mature T cell malignancies enrolled after maximum tolerated dose (MTD) is determined.
- Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide: T-cell Malignancies, Dose Expansion, Arm 2, Dose Level 4
  Arm 2, Dose Level 4: Lenalidomide by oral intake at maximum tolerated dose (MTD) Day 1-10 (7 days lead in for first cycle); CC-486 (5azacitidine) 300 mg by mouth (PO Day) 1 to 10; Romidepsin 12 mg/m^2 intravenous (IV) Day 1 and day 10; Dexamethasone 40 mg PO Day 1 and day 10. Relapsed/refractory mature T cell malignancies enrolled after maximum tolerated dose (MTD) is determined.
- Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide: T-cell Malignancies, Dose Expansion, Arm 3, Dose Level 4
  Arm 3, Dose Level 4: Lenalidomide 20 mg maximum tolerated dose (MTD) by oral intake at on days -7 to 10 of each 21-day cycle (max 6 cycles) with CC-486 (5-azacitidine) at 300mg/day by oral intake on days 1-10, Romidepsin at 12 mg/m^2 by intravenous (IV) infusion on Day 1 and day 10; and Dexamethasone at 40 mg by oral intake on days 1 and 10 of each cycle. Relapsed/refractory mature T cell malignancies enrolled after maximum tolerated dose (MTD) is determined.
- Dose Level -2 Lenalidomide: No participants were enrolled on this dose level. Dose Level-2: Lenalidomide 0 mg Day 1-10 (7 days lead in for first cycle); CC-486 (5azacitidine) 200 mg by mouth (PO Day) 1 to 10; Romidepsin 10 mg/m^2 intravenous (IV) Day 1 and day 10; Dexamethasone 40 mg PO Day 1 and day 10.
Period: Dose Escalation
Arm/Group | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 3 Dose Escalation | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Dose Level -2 Lenalidomide
Started | 2 | 6 | 6 | 3 | 3 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Not Completed | 1 | 5 | 4 | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 3 | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Refused further treatment | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Expansion
Arm/Group | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 3 Dose Escalation | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Dose Level -2 Lenalidomide
Started | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide: T-cell Malignancies, Dose Escalation, Arm 1, Dose Level -1 Arm 1, Dose Level-1: Lenalidomide 2.5 mg Day 1-10 (7 days lead in for first cycle); CC-486 (5azacitidine) 200 mg by mouth (PO Day) 1 to 10; Romidepsin 12 mg/m^2 intravenous (IV) Day 1 and day 10; Dexamethasone 40 mg PO Day 1 and day 10. Relapsed/refractory mature T cell malignancies for determination of maximum tolerated dose (MTD).
- Total: Total of all reporting groups
Arm/Group | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 3 Dose Escalation | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Total
Number analyzed (Participants) | 2 | 6 | 6 | 3 | 3 | 2 | 1 | 3 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5 | 3 | 3 | 1 | 1 | 1 | 19
  >=65 years | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (15.56) | 63.17 (11.46) | 55.67 (8.07) | 46.33 (14.19) | 46.67 (16.29) | 66.5 (9.19) | 65 (0) | 62.67 (21.73) | 58 (13.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 7
  Male | 1 | 4 | 4 | 2 | 3 | 1 | 1 | 3 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 2 | 0 | 1 | 0 | 1 | 10
  White | 0 | 2 | 2 | 1 | 2 | 1 | 0 | 0 | 8
  More Than One Race | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Race Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 2 | 5 | 6 | 3 | 2 | 2 | 1 | 2 | 23
  Ethnicity Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 6 | 6 | 3 | 3 | 2 | 1 | 3 | 26

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD is the dose level at which no more than 1 of up to 6 participants experience dose-limiting toxicity (DLT) during the DLT evaluation window(s), or the dose below that at which at least 2 (of ≤6) participants have DLT. A DLT is defined as any treatment-emergent and related severe (grade ≥3) toxicity related to lenalidomide, romidepsin and/or CC-486 (5-azacitidine) and occurring during the maximum tolerated dose (MTD) observation time, defined as day -7 until end of cycle 1 (normally day 22).
Time Frame: 21 days
Measure: Number; unit: mg/day
Groups:
- All Participants: All participants who completed at least one cycle (21 days) of treatment.
Arm/Group | All Participants
Number analyzed (Participants) | 26
mg/day | 20

2. Primary Outcome: Rate and Severity of Serious and/or Non-serious Adverse Events (AE's) by Grade and Type of Toxicity
Description: Rate and severity of AEs will be summarized by grade and type of toxicity. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: 6 cycles (each cycle is 28 days)
Measure: Number; unit: adverse events
Groups:
- Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide - Serious AE's: Arm 1, Cohort 1, Dose Level -1: Serious AE's
- Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide - Non-Serious AE's: Arm 1, Cohort 1, Dose Level -1: Non-Serious AE's
- Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide - Serious AE's: Arm 1, Cohort 1, Dose Level 1: Serious AE's
- Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide - Non-Serious AE's: Arm 1, Cohort 1, Dose Level 1: Non-Serious AE's
- Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide - Serious AE's: Arm 1, Cohort 1, Dose Level 2: Serious AE's
- Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide - Non-Serious AE's: Arm 1, Cohort 1, Dose Level 2: Non-Serious AE's
- Arm 1, Cohort 1, Dose Level 3 Dose Escalation - Serious AE's: Arm 1, Cohort 1, Dose Level 3: Serious AE's
- Arm 1, Cohort 1, Dose Level 3 Dose Escalation - Non-Serious AE's: Arm 1, Cohort 1, Dose Level 3: Non-Serious AE's
- Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide - Serious AE's: Arm 1, Cohort 1, Dose Level 4: Serious AE's
- Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide - Non-Serious AE's: Arm 1, Cohort 1, Dose Level 4: Non-Serious AE's
- Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide - Serious AE's: Arm 2, Cohort 2, Dose Level 2: Serious AE's
- Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide - Non-Serious AE's: Arm 2, Cohort 2, Dose Level 2: Non-Serious AE's
- Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide - Serious AE's: Arm 2, Cohort 2, Dose Level 4: Serious AE's
- Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide - Non-Serious AE's: Arm 2, Cohort 2, Dose Level 4: Non-Serious AE's
- Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide - Serious AE's: Arm 3, Cohort 2, Dose Level 4: Serious AE's
- Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide - Non-Serious AE's: Arm 3, Cohort 2, Dose Level 4: Non-Serious AE's
Arm/Group | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide - Serious AE's | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide - Non-Serious AE's | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide - Serious AE's | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide - Non-Serious AE's | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide - Serious AE's | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide - Non-Serious AE's | Arm 1, Cohort 1, Dose Level 3 Dose Escalation - Serious AE's | Arm 1, Cohort 1, Dose Level 3 Dose Escalation - Non-Serious AE's | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide - Serious AE's | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide - Non-Serious AE's | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide - Serious AE's | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide - Non-Serious AE's | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide - Serious AE's | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide - Non-Serious AE's | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide - Serious AE's | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide - Non-Serious AE's
Number analyzed (Participants) | 2 | 2 | 6 | 6 | 6 | 6 | 3 | 3 | 3 | 3 | 2 | 2 | 1 | 1 | 3 | 3
adverse events
  Grade 1 Heart failure | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 1 Hypotension | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Fatigue | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 4 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Nausea | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 6 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Vomiting | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Neoplasms benign, malignant&unspecified(incl cysts&polyps)Other specify tumor flare reaction | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Pain in extremity | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Anemia | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 7 | 0 | 6 | 0 | 3 | 0 | 0 | 0 | 0
  Grade 3 Anorexia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Atrial fibrillation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Adrenal insufficiency | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Blood bilirubin increased | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hepatobiliary disorders - Other specify, Drug-Induced liver injury | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Rhabdomyolysis | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Adrenal insufficiency | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Treatment Emergent Grades 3, 4 and/or 5 Adverse Events Possibly Related to Drug Grouped by Severity
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: 6 cycles (each cycle is 28 days)
Measure: Number; unit: adverse events
Arm/Group | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 3 Dose Escalation | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide
Number analyzed (Participants) | 2 | 6 | 6 | 3 | 3 | 2 | 1 | 3
adverse events
  Grade 3 | 13 | 9 | 0 | 4 | 1 | 4 | 1 | 4
  Grade 4 | 4 | 2 | 0 | 4 | 1 | 4 | 0 | 3
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Arm 1, Cohort 1, Dose Level -1, 1, and 2 Treatment Emergent Serious Grades 3, 4, and/or 5 Adverse Events Possibly Related to Drug Grouped by Relationship to the Study Drug and/or Combination
Description: Treatment emergent grades 3, 4, and/or 5 adverse events possibly related grouped by relationship to the study drug (e.g., lenalidomide, romidepsin, CC-486 (5-azacitidine) in any combinations) assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 3 is severe. Grade 4 is life threatening. Grade 5 is death related to adverse event.
Time Frame: 6 cycles (each cycle is 28 days)
Measure: Number; unit: adverse events
Groups:
- Arm 1, Cohort 1, Dose Level -1 Dose Escalation Related to Lenalidomide: Arm 1, Cohort 1, Dose Level -1: adverse events possibly related to lenalidomide.
- Arm 1, Cohort 1, Dose Level -1 - Dose Escalation Related to Romidepsin: Arm 1, Cohort 1, Dose Level -1: adverse events possibly related to romidepsin.
- Arm 1, Cohort 1, Dose Level -1 - Dose Escalation Related to CC-486 (5-azacitidine): Arm 1, Cohort 1, Dose Level -1: adverse events possibly related to CC-486 (5-azacitidine).
- Arm 1, Cohort 1, Dose Level -1: Dose Escalation Related to Any Combination: Arm 1, Cohort 1, Dose Level -1: adverse events possibly related to any combination.
- Arm 1, Cohort 1, Dose Level 1 - Dose Expansion Related to Lenalidomide: Arm 1, Cohort 1, Dose Level 1: adverse events possibly related to lenalidomide.
- Arm 1, Cohort 1, Dose Level 1 - Dose Expansion Related to Romidepsin: Arm 1, Cohort 1, Dose Level 1: adverse events possibly related to romidepsin.
- Arm 1, Cohort 1, Dose Level 1 - Dose Expansion Related to CC-486 (5-azacitidine): Arm 1, Cohort 1, Dose Level 1: adverse events possibly related to CC-486 (5-azacitidine).
- Arm 1, Cohort 1, Dose Level 1 - Dose Expansion Related to Any Combination: Arm 1, Cohort 1, Dose Level 1: adverse events possibly related to any combination.
- Arm 1, Cohort 1, Dose Level 2 - Dose Escalation Related to Lenalidomide: Arm 1, Cohort 1, Dose Level 2: adverse events possibly related to lenalidomide.
- Arm 1, Cohort 1, Dose Level 2 - Dose Escalation Related to Romidepsin: Arm 1, Cohort 1, Dose Level 2: adverse events possibly related to romidepsin.
- Arm 1, Cohort 1, Dose Level 2 - Dose Escalation Related to CC-486 (5-azacitidine): Arm 1, Cohort 1, Dose Level 2: adverse events possibly related to CC-486 (5-azacitidine).
- Arm 1, Cohort 1, Dose Level 2 - Dose Escalation Related to Any Combination: Arm 1, Cohort 1, Dose Level 2: adverse events possibly related to any combination.
Arm/Group | Arm 1, Cohort 1, Dose Level -1 Dose Escalation Related to Lenalidomide | Arm 1, Cohort 1, Dose Level -1 - Dose Escalation Related to Romidepsin | Arm 1, Cohort 1, Dose Level -1 - Dose Escalation Related to CC-486 (5-azacitidine) | Arm 1, Cohort 1, Dose Level -1: Dose Escalation Related to Any Combination | Arm 1, Cohort 1, Dose Level 1 - Dose Expansion Related to Lenalidomide | Arm 1, Cohort 1, Dose Level 1 - Dose Expansion Related to Romidepsin | Arm 1, Cohort 1, Dose Level 1 - Dose Expansion Related to CC-486 (5-azacitidine) | Arm 1, Cohort 1, Dose Level 1 - Dose Expansion Related to Any Combination | Arm 1, Cohort 1, Dose Level 2 - Dose Escalation Related to Lenalidomide | Arm 1, Cohort 1, Dose Level 2 - Dose Escalation Related to Romidepsin | Arm 1, Cohort 1, Dose Level 2 - Dose Escalation Related to CC-486 (5-azacitidine) | Arm 1, Cohort 1, Dose Level 2 - Dose Escalation Related to Any Combination
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
adverse events
  Grade 3 Serious Anorexia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Serious Atrial fibrillation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 or 5 Any Serious Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Anemia | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Lymphocyte count decreased | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Platelet count decreased | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Ejection fraction decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Hypokalemia | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Neutrophil count decreased | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4 | 1 | 1 | 1 | 1
  Grade 3 Non-Serious Platelet count decreased | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 1 | 0 | 0 | 1
  Grade 3 Non-serious White blood cell decreased | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Fatigue | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
  Grade 3 Non-serious Weight loss | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Grade 4 Non-serious Platelet count decreased | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 4 Non-serious Neutrophil count decreased | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0
  Grade 4 White blood cell decreased | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0

5. Primary Outcome: Arm 1, Cohort 1, Dose Level 3, and Arm 1, Cohort 1, Dose Level 4 Treatment Emergent Serious Grades 3, 4, and/or 5 Adverse Events Possibly Related to Drug Grouped by Relationship to the Study Drug and/or Combination
Description: as for outcome 4
Time Frame: 6 cycles (each cycle is 28 days)
Measure: Number; unit: adverse events
Groups:
- Arm 1, Cohort 1, Dose Level 3 Dose Escalation Related to Lenalidomide: Arm 1, Cohort 1, Dose Level 3: adverse events possibly related to lenalidomide.
- Arm 1, Cohort 1, Dose Level 3 - Dose Escalation Related to Romidepsin: Arm 1, Cohort 1, Dose Level 3: adverse events possibly related to romidepsin.
- Arm 1, Cohort 1, Dose Level 3 - Dose Escalation Related to CC-486 (5-azacitidine): Arm 1, Cohort 1, Dose Level 3: adverse events possibly related to CC-486 (5-azacitidine).
- Arm 1, Cohort 1, Dose Level 3: Dose Escalation Related to Any Combination: Arm 1, Cohort 1, Dose Level 3: adverse events possibly related to any combination.
- Arm 1, Cohort 1, Dose Level 4 - Dose Escalation Related to Lenalidomide: Arm 1, Cohort 1, Dose Level 4: adverse events possibly related to lenalidomide.
- Arm 1, Cohort 1, Dose Level 4 - Dose Escalation Related to Romidepsin: Arm 1, Cohort 1, Dose Level 4: adverse events possibly related to romidepsin.
- Arm 1, Cohort 1, Dose Level 4 - Dose Escalation Related to CC-486 (5-azacitidine): Arm 1, Cohort 1, Dose Level 4: adverse events possibly related to CC-486 (5-azacitidine).
- Arm 1, Cohort 1, Dose Level 4 - Dose Escalation Related to Any Combination: Arm 1, Cohort 1, Dose Level 4: adverse events possibly related to any combination.
Arm/Group | Arm 1, Cohort 1, Dose Level 3 Dose Escalation Related to Lenalidomide | Arm 1, Cohort 1, Dose Level 3 - Dose Escalation Related to Romidepsin | Arm 1, Cohort 1, Dose Level 3 - Dose Escalation Related to CC-486 (5-azacitidine) | Arm 1, Cohort 1, Dose Level 3: Dose Escalation Related to Any Combination | Arm 1, Cohort 1, Dose Level 4 - Dose Escalation Related to Lenalidomide | Arm 1, Cohort 1, Dose Level 4 - Dose Escalation Related to Romidepsin | Arm 1, Cohort 1, Dose Level 4 - Dose Escalation Related to CC-486 (5-azacitidine) | Arm 1, Cohort 1, Dose Level 4 - Dose Escalation Related to Any Combination
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
adverse events
  Grade 3 Serious Blood bilirubin increased | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Serious Hepatobiliary disorders - Other specify, Drug-Induced liver injury | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Serious Rhabdomyolysis | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 0
  Any Grade 4 and/or 5 Serious Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Acute kidney injury | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Alanine aminotransferase increased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Anemia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Aspartate aminotransferase increased | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Blood bilirubin increased | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Non-serious CPK increased | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Fatigue | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Hypotension | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Lymphocyte count decreased | 4 | 4 | 4 | 4 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Neutrophil count decreased | 3 | 3 | 3 | 3 | 2 | 2 | 2 | 2
  Grade 3 Platelet count decreased | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 White blood cell decreased | 3 | 3 | 0 | 0 | 1 | 1 | 1 | 1
  Grade 4 CPK increased | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Grade 4 Lymphocyte count decreased | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2

6. Primary Outcome: Arm 2, Cohort 2, Dose Level 2 and 4; and Arm 3, Cohort 2, Dose Level 4 Treatment Emergent Serious Grades 3, 4, and/or 5 Adverse Events Possibly Related to Drug Grouped by Relationship to the Study Drug and/or Combination
Description: as for outcome 4
Time Frame: 6 cycles (each cycle is 28 days)
Measure: Number; unit: adverse events
Groups:
- Arm 2, Cohort 2, Dose Level 2 - Dose Expansion Related to Lenalidomide: Arm 2, Cohort 2, Dose Level 2: adverse events possibly related to lenalidomide.
- Arm 2, Cohort 2, Dose Level 2 - Dose Expansion Related to Romidepsin: Arm 2, Cohort 2, Dose Level 2: adverse events possibly related to romidepsin.
- Arm 2, Cohort 2, Dose Level 2 - Dose Expansion Related to CC-486 (5-azacitidine): Arm 2, Cohort 2, Dose Level 2: adverse events possibly related to CC-486 (5-azacitidine).
- Arm 2, Cohort 2, Dose Level 2 - Dose Expansion Related to Any Combination: Arm 2, Cohort 2, Dose Level 2: adverse events possibly related to any combination.
- Arm 2, Cohort 2, Dose Level 4 - Dose Expansion Related to Lenalidomide: Arm 2, Cohort 2, Dose Level 4: adverse events possibly related to lenalidomide.
- Arm 2, Cohort 2, Dose Level 4 - Dose Expansion Related to Romidepsin: Arm 2, Cohort 2, Dose Level 4: adverse events possibly related to romidepsin.
- Arm 2, Cohort 2, Dose Level 4 - Dose Expansion Related to CC-486 (5-azacitidine): Arm 2, Cohort 2, Dose Level 4: adverse events possibly related to CC-486 (5-azacitidine).
- Arm 2, Cohort 2, Dose Level 4 - Dose Expansion Related to Any Combination: Arm 2, Cohort 2, Dose Level 4: adverse events possibly related to any combination.
- Arm 3, Cohort 2, Dose Level 4 - Dose Expansion Related to Lenalidomide: Arm 3, Cohort 2, Dose Level 4: adverse events possibly related to lenalidomide.
- Arm 3, Cohort 2, Dose Level 4 - Dose Expansion Related to Romidepsin: Arm 3, Cohort 2, Dose Level 4: adverse events possibly related to romidepsin.
- Arm 3, Cohort 2, Dose Level 4 - Dose Expansion Related to CC-486 (5-azacitidine): Arm 3, Cohort 2, Dose Level 4: adverse events possibly related to CC-486 (5-azacitidine).
- Arm 3, Cohort 2, Dose Level 4 - Dose Expansion Related to Any Combination: Arm 3, Cohort 2, Dose Level 4: adverse events possibly related to any combination.
Arm/Group | Arm 2, Cohort 2, Dose Level 2 - Dose Expansion Related to Lenalidomide | Arm 2, Cohort 2, Dose Level 2 - Dose Expansion Related to Romidepsin | Arm 2, Cohort 2, Dose Level 2 - Dose Expansion Related to CC-486 (5-azacitidine) | Arm 2, Cohort 2, Dose Level 2 - Dose Expansion Related to Any Combination | Arm 2, Cohort 2, Dose Level 4 - Dose Expansion Related to Lenalidomide | Arm 2, Cohort 2, Dose Level 4 - Dose Expansion Related to Romidepsin | Arm 2, Cohort 2, Dose Level 4 - Dose Expansion Related to CC-486 (5-azacitidine) | Arm 2, Cohort 2, Dose Level 4 - Dose Expansion Related to Any Combination | Arm 3, Cohort 2, Dose Level 4 - Dose Expansion Related to Lenalidomide | Arm 3, Cohort 2, Dose Level 4 - Dose Expansion Related to Romidepsin | Arm 3, Cohort 2, Dose Level 4 - Dose Expansion Related to CC-486 (5-azacitidine) | Arm 3, Cohort 2, Dose Level 4 - Dose Expansion Related to Any Combination
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 3 | 3 | 3 | 3
adverse events
  Any Grade 3, 4, and/or 5 Serious Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Anemia | 1 | 1 | 1 | 1 | 7 | 7 | 7 | 7 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Anorexia | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Non-serious Hypokalemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Platelet count decreased | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4 | 0 | 0 | 0 | 0
  Grade 4 Neutrophil count decreased | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 4 Platelet count decreased | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0

7. Secondary Outcome: Overall Response Rate (Complete Response + Partial Response)
Description: The response rate will be estimated using the Kaplan-Meier curve and reported along with a 95% confidence interval. Response was measured by the Response Evaluation Criteria in Lymphoma (RECIL) 2017 criteria. Complete response (CR) is disappearance of all target lesions and all nodes with long axis <10mm. Partial response (PR) is a ≥30% decrease in the sum of longest diameters of target lesions but not a CR.
Time Frame: 6 cycles (each cycle is 28 days)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 3 Dose Escalation | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide
Number analyzed (Participants) | 2 | 6 | 6 | 3 | 3 | 2 | 1 | 3
percentage of participants
  Complete Response | 50 [47.3 to 52.7] | 16.6 [15.3 to 18.0] | 33.3 [31.8 to 34.8] | 66 [64.0 to 68.0] | 100 [98 to 100] | 50 [47.3 to 52.7] | 100 [100 to 100] | 100 [97.3 to 100]
  Partial Response | 50 [47.3 to 52.7] | 0 [0 to 0] | 33.3 [31.8 to 34.8] | 66 [64.0 to 68.0] | 100 [98 to 100] | 50 [47.3 to 52.7] | 0 [0 to 0] | 50 [47.3 to 52.7]

8. Secondary Outcome: Progression-free Survival (PFS) in Months Reported Along With a 95% Confidence Interval
Description: PFS will be estimated using the Kaplan-Meier curve and reported along with a 95% confidence interval. PFS is defined as the duration of time from the date of study enrollment until time of disease relapse, disease progression, or death, whichever occurs first measured by the Response Evaluation Criteria in Lymphoma (RECIL) 2017 criteria. Progressive disease is >20% increase in the sum of longest diameters of target lesions. Disease relapse is defined as new areas of disease or >50% increase in growth of target lesion.
Time Frame: up to a median of 13.1 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 3 Dose Escalation | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide
Number analyzed (Participants) | 2 | 6 | 6 | 3 | 3 | 2 | 1 | 3
Months | 5.3 [4.8 to 5.8] | 1.7 [1.4 to 2.0] | NA [NA to NA] — The median was not reached as there were not enough events. | 3.7 [3.1 to 4.3] | 9.2 [8.6 to 10.0] | 3.6 [3.3 to 3.9] | 13.1 [13.1 to 13.1] | 3.4 [3.0 to 3.8]

9. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR will be estimated using the Kaplan-Meier curve and reported along with a 95% confidence interval. Response was measured by the Response Evaluation Criteria in Lymphoma (RECIL) 2017 criteria. Complete response (CR) is disappearance of all target lesions and all nodes with long axis <10mm.
Time Frame: 6 cycles (each cycle is 28 days)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 3 Dose Escalation | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide
Number analyzed (Participants) | 2 | 6 | 6 | 3 | 3 | 2 | 1 | 3
percentage of participants | 0 [0 to 0] | 16.6 [15.3 to 18.0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 100 [100 to 100] | 50 [47.3 to 52.7]

10. Secondary Outcome: Duration of Response (DOR) in Months Reported Along With a 95% Confidence Interval
Description: DOR will be determined and reported along with a 95% confidence interval. DOR is measured from the time measurement criteria are met for complete response (CR) or partial response (PR (whichever is recorded first) until the first date that recurrent or progressive disease is objectively documented. Response was measured by the Response Evaluation Criteria in Lymphoma (RECIL) 2017 criteria. Complete response (CR) is disappearance of all target lesions and all nodes with long axis <10mm. Partial response (PR) is a ≥30% decrease in the sum of longest diameters of target lesions but not a CR. Progressive disease is >20% increase in the sum of longest diameters of target lesions.
Time Frame: up to a median of 11.7 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 3 Dose Escalation | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide
Number analyzed (Participants) | 2 | 6 | 6 | 3 | 3 | 2 | 1 | 3
Months | 5.8 [5.2 to 6.4] | NA [NA to NA] — The median was not reached as there were not enough events. | NA [NA to NA] — The median was not reached as there were not enough events. | 2.1 [1.8 to 2.4] | 6.0 [5.7 to 6.3] | 3.4 [3.0 to 3.8] | 11.7 [11.7 to 11.7] | 1.5 [1.1 to 1.9]

11. Secondary Outcome: Overall Survival (OS)
Description: OS will be estimated using the Kaplan-Meier curve and reported along with a 95% confidence interval. OS is defined as the time from the date of study enrollment until time of death from any cause.
Time Frame: up to a median of 8.7 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 3 Dose Escalation | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide
Number analyzed (Participants) | 2 | 6 | 6 | 3 | 3 | 2 | 1 | 3
Months | 8.7 [8.1 to 9.3] | 4.6 [4.2 to 5.0] | NA [NA to NA] — The median was not reached as there were not enough events. | NA [NA to NA] — The median was not reached as there were not enough events. | NA [NA to NA] — The median was not reached as there were not enough events. | 4.5 [3.9 to 5.1] | NA [NA to NA] — The median was not reached as there were not enough events. | NA [NA to NA] — The median was not reached as there were not enough events.

12. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 3 Dose Escalation | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide
Number analyzed (Participants) | 2 | 6 | 6 | 3 | 3 | 2 | 1 | 3
Participants | 2 | 6 | 6 | 3 | 3 | 2 | 1 | 3

13. Other Pre Specified Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: A DLT is defined as any treatment-emergent and related severe (grade ≥3) toxicity related to lenalidomide, romidepsin and/or CC-486 (5-azacitidine) and occurring during the maximum tolerated dose (MTD) observation time, defined as day -7 until end of cycle 1 (normally day 22). Grade 4 is life threatening, and Grade 5 is death related to adverse event. Serious toxicity was assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Time Frame: Day -7 until end of cycle 1 (normally day 22)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 3 Dose Escalation | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide
Number analyzed (Participants) | 2 | 6 | 6 | 3 | 3 | 2 | 1 | 3
Participants
  Grade 3 | 0 | 0 | 0 | 00 | 0 | 0 | 0 | 0
  Grade 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed at a median follow-up of 20.4 months. Adverse Events was monitored/assessed from the first study intervention, Study Day 1 through 30 days after the last intervention, or disease progression, up to 3.5 years.
Arm/Group | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide | Arm 1, Cohort 1, Dose Level 3 Dose Escalation | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide
All-Cause Mortality (participants affected / at risk) | 2/2 | 3/6 | 3/6 | 1/3 | 0/3 | 1/2 | 1/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/6 | 1/6 | 2/3 | 0/3 | 0/2 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 6/6 | 6/6 | 3/3 | 3/3 | 2/2 | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide (N=2) | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide (N=6) | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide (N=6) | Arm 1, Cohort 1, Dose Level 3 Dose Escalation (N=3) | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide (N=3) | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide (N=2) | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide (N=1) | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide (N=3)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify: Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — (incl cysts and polyps) - Other, specify: Tumor flare reaction
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1, Cohort 1, Dose Level -1, Dose Escalation Lenalidomide (N=2) | Arm 1, Cohort 1, Dose Level 1, Dose Expansion Lenalidomide (N=6) | Arm 1, Cohort 1, Dose Level 2, Dose Escalation Lenalidomide (N=6) | Arm 1, Cohort 1, Dose Level 3 Dose Escalation (N=3) | Arm 1, Cohort 1, Dose Level 4, Dose Escalation Lenalidomide (N=3) | Arm 2, Cohort 2, Dose Level 2, Dose Expansion Lenalidomide (N=2) | Arm 2, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide (N=1) | Arm 3, Cohort 2, Dose Level 4, Dose Expansion Lenalidomide (N=3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (2) | 0 (0) | 1 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (10) | 4 (16) | 4 (10) | 3 (14) | 2 (3) | 2 (5) | 1 (18) | 1 (5)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (4) | 1 (1) | 1 (9) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify: low iron level (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (4) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (6) | 1 (4) | 2 (4) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 3 (4) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Eye disorders - Other, specify: Corneal Thinning (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify: Itchy eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify: Light Sensitivity (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify: double vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (3) | 2 (2) | 4 (7) | 1 (2) | 2 (6) | 1 (1) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 3 (9) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: Increased thirst, Intermittent (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (6) | 2 (2) | 1 (1) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (14) | 1 (3) | 3 (4) | 2 (3) | 0 (0) | 1 (4) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify: Decreased iron (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (11) | 0 (0) | 1 (2) | 3 (21) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: Fracture, compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (5) | 4 (5) | 1 (1) | 3 (8) | 1 (1) | 0 (0) | 1 (2)
Nervous system disorders - Other, specify: Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 5 (25) | 5 (12) | 2 (11) | 1 (7) | 0 (0) | 1 (2) | 1 (2)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (19) | 5 (23) | 4 (12) | 2 (10) | 2 (2) | 0 (0) | 1 (14) | 2 (12)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (3) | 2 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 3 (7) | 3 (7) | 1 (1) | 2 (5) | 1 (1) | 0 (0) | 1 (1)
Vulval infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (1) | 2 (3) | 2 (6) | 3 (10) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (4) | 1 (3) | 2 (10) | 3 (6) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT04447027/Prot_SAP_002.pdf
  • Informed Consent Form (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT04447027/ICF_001.pdf